CLINICAL TRIAL: NCT04137367
Title: A Personalized Approach to Effects of Affective Bias Modification on Symptom Change and Rumination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Extrastiftelsen (Other); Diakonhjemmet Hospital (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Nils Inge Landrø, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/FO249225
Record Dates: First submitted 2019-10-10; First posted 2019-10-24 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
Keywords: Rumination; Attention bias modification; Transdiagnostic
MeSH Terms: conditions — Depressive Disorder, Major; Rumination Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Affective Bias Modification (Experimental): Computer based Affective Bias Modification
  Interventions: Behavioral: Affective bias modification
- Sham Affective Bias Modification (Sham Comparator): Computer based sham Affective Bias Modification
  Interventions: Behavioral: Sham Affective bias modification
- Assesment only (No Intervention): Only assessments are conducted

INTERVENTIONS:
Behavioral: Affective bias modification — In the Affective bias modification (ABM) procedure, paired stimuli (e.g. a negative and a positive facial expression) are presented on a laptop screen, followed by one or two probes (dots) appearing in the spatial location of one of the stimuli. Participants are then required to press one of two buttons as quickly as possible to indicate the number of dots in the probe. Stimuli presentation time is 50% 500 ms and 50 % 1000 ms (evenly distributed throughout the task). In total, the ABM will comprise 90 trials of paired images of faces of different valences. In the active condition, the probe appears at the location of the most positive stimuli of each pair in 87 % of trials (encouraging a positive affective bias). Participants will do ABM in their homes (approx. 5 min.) twice a day for two weeks (28 sessions) using laptop computers provided by us.
  Other Names: Attention Bias Modification
  Arms: Active Affective Bias Modification
Behavioral: Sham Affective bias modification — In the Affective bias modification (ABM) procedure, paired stimuli (e.g. a negative and a positive facial expression) are presented on a laptop screen, followed by one or two probes (dots) appearing in the spatial location of one of the stimuli. Participants are then required to press one of two buttons as quickly as possible to indicate the number of dots in the probe. Stimuli presentation time is 50% 500 ms and 50 % 1000 ms (evenly distributed throughout the task). In total, the ABM will comprise 90 trials of paired images of faces of different valences. In the sham condition, the probe appears at the location of the most positive stimuli of each pair in 50 % of trials (no contingency between facial expressions shown and the probe location). Participants will do ABM in their homes (approx. 5 min.) twice a day for two weeks (28 sessions) using laptop computers provided by us.
  Other Names: Sham Attention bias modification
  Arms: Sham Affective Bias Modification

SUMMARY:
This study evaluates the effect of a computerized intervention for depressive symptoms called Affective Bias Modification (ABM). A third of the patients will receive active ABM, a third will receive sham ABM and a third will undergo assessment only. The study will investigate if rumination mediates the effect of the intervention and investigate if specific symptom profiles affect the effect of the intervention.

DETAILED DESCRIPTION:
A main aim of the project is to investigate how the effects of an ABM intervention on depressive symptoms are mediated by transdiagnostic rumination and how characteristics of the symptom network moderate these effects. The Affective Bias Modification Task (ABM) will be applied in a randomized controlled, double blind clinical trial with 6 months follow-up. Personalized networks are generated from prospective assessment of depression-related processes at baseline and follow-ups. Patients (n = 150) will be recruited from out-patient clinics at Diakonhjemmet Hospital, and randomized into one of three conditions: active, sham and assessment only. Patients aged 18-65 with depression (major depressive disorder) or bipolar disorder 2, with or without comorbid anxiety and/or alcohol use disorder will be included. The main hypothesis is that subjects who are in the active ABM group will exhibit less tendency for stress related (state) rumination compared to those in the placebo group. Active vs placebo ABM will decrease depressive symptoms (6 months) and this effect will be mediated by the change in state rumination. Densely connected symptom network and high strength centrality of rumination at baseline will moderate the effect of ABM. By combining mechanisms research with a personalized symptom network approach, this study will be in the forefront of understanding how a drug-free treatment option works and for whom it works best.

ELIGIBILITY:
Inclusion Criteria:

- Current or remitted Major Depressive Disorder, with or without anxiety, with or without alcohol use disorder

Exclusion Criteria:

* Neurological disorder, mania, and/or psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Inge Landrø, Dr.Philos, Principal Investigator — University of Oslo
Locations (1):
- Department of Psychology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bo R, Kraft B, Joormann J, Jonassen R, Harmer CJ, Landro NI. Cognitive predictors of stress-induced mood malleability in depression. Anxiety Stress Coping. 2024 Mar;37(2):278-292. doi: 10.1080/10615806.2023.2255531. Epub 2023 Sep 11. PMID 37695740
- [Derived] Bo R, Kraft B, Pedersen ML, Joormann J, Jonassen R, Osnes K, Harmer CJ, Landro NI. The effect of attention bias modification on depressive symptoms in a comorbid sample: a randomized controlled trial. Psychol Med. 2023 Oct;53(13):6389-6396. doi: 10.1017/S0033291722003956. Epub 2023 Jan 9. PMID 36617964
- See also: Project web page — https://www.sv.uio.no/psi/english/research/projects/affective-bias-modification/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between Nov 19, 2019, and Aug 17, 2021 using local advertisements and social media. Entrance to the trial was via self-referral by phone or online registration.
Pre-assignment Details: Did not meet the inclusion criteria (N=4), Declined to participate (n=4), Not able to get in contact with (N=4).
Groups:
- Assessment Only: Only assessments were conducted.
Period: Overall Study
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assessment Only
Started | 50 | 51 | 7
Completed | 42 | 45 | 3
Not Completed | 8 | 6 | 4
Not completed — Lost to Follow-up | 8 | 6 | 4

BASELINE CHARACTERISTICS:
Population: 16 persons withdrew before baseline assessment.
Groups:
- Assesment Only: No intervention.
- Total: Total of all reporting groups
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assesment Only | Total
Number analyzed (Participants) | 42 | 45 | 5 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Technical problems led to missing data for two participant.
  years
    number analyzed (Participants) | 41 | 45 | 4 | 90
    (all) | 44.3 (10.4) | 43.2 (11.6) | 36.8 (18.2) | 43.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 3 | 67
  Male | 14 | 9 | 2 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 42 | 45 | 5 | 92
Education level (ISCED) [Mean (Standard Deviation); unit: units on a scale] — International Standard Classification of Education (ISCED), min=0, max=8, value represents average education level for the group. Higher score means higher education.
  ISCED 0: Early childhood education ('less than primary' for educational attainment) ISCED 1: Primary education ISCED 2: Lower secondary education ISCED 3: Upper secondary education ISCED 4: Post-secondary non-tertiary education ISCED 5: Short-cycle tertiary education ISCED 6: Bachelor's or equivalent level ISCED 7: Master's or equivalent level ISCED 8: Doctoral or equivalent level Population: Technical problems led to missing data for two participants.
  units on a scale
    number analyzed (Participants) | 41 | 45 | 4 | 90
    (all) | 5.7 (1.3) | 5.8 (1.2) | 4.8 (2.1) | 5.7 (1.3)
Beck's Depression Inventory (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — Becks Depression Inventory-II (BDI-II) Self-report scale including 21 items. Likert scale 0-3. Higher scores represent more severe depression symptoms. Min = 0, Max = 63. The presented value is the average total score per group. Population: Technical problems led to missing data for two participants.
  units on a scale
    number analyzed (Participants) | 41 | 45 | 4 | 90
    (all) | 23.1 (10.6) | 26.3 (9.8) | 18.2 (3.8) | 24.4 (9.9)
Beck's Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — Self-report scale including 19 items. Likert scale 0-3. Min = 0, Max = 57. The average total score per group is reported. Higher scores represent more severe anxiety symptoms. Population: Technical problems led to missing data for one participant.
  units on a scale
    number analyzed (Participants) | 41 | 45 | 5 | 91
    (all) | 13.1 (8.8) | 16.2 (8.9) | 12.0 (7.5) | 14.6 (8.8)
Alcohol Use Disorder Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — Self-report scale including 9 items. Likert scale 0-4. Min = 0, Max = 36. The average total score per groups is reported. Higher scores implies increased risk of alcohol use disorder. Population: Technical problems led to missing data for one participant.
  units on a scale
    number analyzed (Participants) | 41 | 45 | 5 | 91
    (all) | 5.8 (4.7) | 5.5 (5.6) | 3.6 (5.5) | 5.5 (5.6)
Brief State Rumination Inventory (BSRI) [Mean (Standard Deviation); unit: units on a scale] — Measures state rumination in response to a stress induction on a 8-item scale on a 0-100 visual analogue scale. The value reported is the total score divided by 8. Min = 0, max = 100.
  Higher values represent more state rumination. Population: Technical problems led to missing data for one participant. Data for this outcome measure was only obtained at baseline and post-intervention, not at 6 months follow-up, as the intention of adopting this measure was to investigate if it mediated the association between the intervention and the primary outcome.
  units on a scale
    number analyzed (Participants) | 41 | 45 | 5 | 91
    (all) | 36.4 (18.7) | 38.3 (17.5) | 22.3 (20.7) | 36.6 (18.4)
Attentional bias [Mean (Standard Deviation); unit: milliseconds] — One session of computerized sham Attentional Bias Modification (ABM), which is based on a dot probe-task, conducted within the lab setting. The value presented is the difference in average reaction time to targets displayed in the location of the previously presented negative stimuli compared to the average reaction time to targets displayed in the location of the relatively more positive (happy-neutral) stimuli, presented in milliseconds. A positive value represents a bias away from negative stimuli, while a negative value represents a bias towards negative. Population: Technical problems led to missing data for one participant. Data for this outcome measure was only obtained at baseline and post-intervention, not at 6 months follow-up, as the intention of adopting this measure was to investigate if the intervention modified its intended mechanism
  milliseconds
    number analyzed (Participants) | 41 | 45 | 5 | 91
    (all) | -10.7 (26.4) | -4.7 (36.0) | -17.1 (29.3) | -8.1 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Depressive Symptoms: Becks Depression Inventory-II
Description: Self-reported depressive symptoms 6 months after the ABM intervention based on a 21-item scale. Each item is scored 0-3 (where scoring description is adapted to each item), yielding a score from 0-63.
Time Frame: At 6 months follow-up
Population: Participants that had baseline and/or outcome data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Assessment Only: No intervention was given, only assessments were conducted.
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assessment Only
Number analyzed (Participants) | 42 | 45 | 5
score on a scale | 19.1 (1.7) | 16.5 (1.6) | 5.3 (5.5)
Statistical Analysis 1: Comparison: Active Affective Bias Modification vs Sham Affective Bias Modification; We estimated a priori that a total of 100 participants would be needed to detect a difference between ABM and sham condition, with a two-tailed α of 0.05 and (1-β) of .80. Power calculation was based on the assumption that 50 % of the participants allocated to ABM would report a minimum of 3 points reduction on BDI-II at six months, compared to 20 % in the sham condition. Assuming 15 % lost to follow up, power calculation indicated the need for 50 participants in each condition; Test type: Other; p = .05, Mixed Models Analysis

2. Primary Outcome: State Rumination: Brief State Rumination Inventory (BSRI)
Description: Change in self-reported state rumination after the stress induction from pre to post intervention on a 8 item scale. Difference score: BSRI post intervention - BRSI Baseline. A negative score means reduction in state rumination over the intervention. Each item is scored on a 0-100 Visual Analogue Scale. The total score divided by 8 to provide the mean item total score, hence the min= 0 and max = 100 for each of the BSRI assessment time points. It was hypothesized that change in state rumination over the intervention period would mediate the effect of ABM on depressive symptoms at six months follow up.
Time Frame: At baseline and two weeks follow up.
Population: 10 persons were lost to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Assesment Only: No intervention was given.
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assesment Only
Number analyzed (Participants) | 37 | 41 | 4
score on a scale | -.7 (13.3) | -5.8 (19.1) | -.8 (7.4)

3. Primary Outcome: State Rumination: Brief State Rumination Inventory
Description: Self-reported state rumination after stress induction on a 8 item scale. Each item is scored on a 0-100 Visual Analogue Scale, yielding a score from 0-800, which is reported divided by 8 to provide a mean total item score. Hence the min= 0 and max = 100. A higher score indicates more state rumination.
Time Frame: At two weeks follow up.
Population: 10 participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Assessment Only: No intervention.
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assessment Only
Number analyzed (Participants) | 37 | 41 | 4
score on a scale | 34.2 (15.8) | 32.3 (15.8) | 23.4 (20.2)

4. Secondary Outcome: Affective Bias: Dot-probe Task
Description: Change in reaction time in milliseconds to probes in the location of the positive facial stimuli compared to probes in the location of the negative stimuli. Positive number implies reduction in negative bias.
Time Frame: From baseline to two weeks follow up
Population: Nine participants were lost to follow up. Technical error led to loss of data on the follow up in the assessment only condition.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assessment Only
Number analyzed (Participants) | 35 | 42 | 0
milliseconds | 18.0 (28.4) | 9.4 (40.3) |

5. Secondary Outcome: Symptom Network Change: Experience Sampling of Depressive Symptoms
Description: Changed centrality of rumination in networks estimated based on a 9-item experience sampling questionnaire of self-reported depressive symptoms scored on a 0-100 visual analogue scale (higher value, more symptoms; reversing interest, positive affect and activity; Kraft et al., 2023, Psychiatry Research Communications). Two person-specific networks (pre and post-intervention) were estimated using the var1-function in the R package psychonetrics, with full-information maximum likelihood estimator, based on the experience sampling questionnaires that were administrated 5 times/day for 14 days before and after the intervention. Centrality of rumination in these networks were calculated using qgraph (Epskamp et al., 2012) and standardized. Change in rumination centrality was calculated as difference between rumination centrality in the two estimated networks, and higher number indicate increased centrality of rumination (post-pre).
Time Frame: From two weeks prior to baseline to two weeks after the two-week intervention.
Population: Pre-processing of ESM-data excluded participants who responded to less than 30 measurements.
Measure: Mean (Standard Deviation); unit: standardized values
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assesment Only
Number analyzed (Participants) | 14 | 16 | 0
standardized values | .0175 (.0819) | -.685 (.789) |

6. Secondary Outcome: Symptom Network: Experience Sampling of Depressive Symptoms
Description: Centrality of rumination in networks based on a 9-item experience sampling questionnaire of self-reported depressive symptoms scored on a 0-100 visual analogue scale (higher value, more symptoms; reversing interest, positive affect and activity; Kraft et al., 2023, Psychiatry Research Communications). Person-specific networks were estimated using the var1-function in the R package psychonetrics, with full-information maximum likelihood estimator, based on the experience sampling questionnaires that were administrated 5 times/day for 14 days after the two-week intervention. Centrality of rumination in this network was calculated using qgraph (Epskamp et al., 2012) and standardized. Higher number indicate higher centrality of rumination.
Time Frame: Two weeks after the two-week intervention.
Population: Participants who responded to 30 measurements or more.
Measure: Mean (Standard Deviation); unit: standardized values
Groups:
- Assessment Only: No intervention was given.
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assessment Only
Number analyzed (Participants) | 22 | 24 | 0
standardized values | .108 (.785) | -.230 (.824) |

ADVERSE EVENTS:
Time Frame: 6 months follow-up after intervention
Description: Participant self-report.
Arm/Group | Active Affective Bias Modification | Sham Affective Bias Modification | Assesment Only
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/7
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04137367/Prot_SAP_000.pdf